CLINICAL TRIAL: NCT04411810
Title: SpotCheck: Comparison of Enhanced Telemedicine Versus In-person Evaluation for the Diagnosis of Skin Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-01242
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants with skin lesions (Experimental): Participants who have up to 3 concerning skin lesions will be evaluated by both an in-person dermatologist and a team of three teledermatologists(board-certified dermatologists). The teledermatoogy team will deliver a consensus recommendation. If either the in-person dermatologist or teledermatologists are concerned that the skin spot(s) may be a skin cancer, a biopsy will be recommended and can be performed at no charge. Or if both agree that the spot(s) are not concerning for skin cancer, no biopsy will be needed.
  Interventions: Device: Nevisense 3.0; Device: Dermlite Cam; Procedure: Skin biopsy; Device: Barco Demetra

INTERVENTIONS:
Device: Nevisense 3.0 — Nevisense, an AI-based point-of-care system for the non-invasive evaluation of irregular moles remains the only FDA approved system available for melanoma detection in the US. Nevisense 3.0 will be used as a one-time exposure of <8 seconds per lesion. Disposable electrodes that contact the participant are 5mm x 5mm in size. Nevisense 3.0 measures electrical impedance of skin lesions and provides an output called the electrical impedence spectroscopy (EIS) score. Electrical impedance is a measure of a material's overall resistance to the flow of alternating electric currents of various frequencies. The principle is that electrical impedance is different in normal versus abnormal tissue.
Device: Dermlite Cam — Dermlite Cam is a digital camera that captures images of the skin under cross-polarized and non-polarized light and is 510(k) exempt. The DermLite Cam device appears as a single piece camera with a charging cable and USB computer cable. As part of the camera unit, an extensor arm exists to allow for the capture of standardized clinical images. The DermLite Cam will be used to acquire 3 images of <5 seconds per lesion (one clinical, one polarized dermoscopic, and one non-polarized dermoscopic). NOTE - for the purposes of this study, teledermatology images (dermoscopic and clinical - at approximately 6 inches, 12 inches, and 18 inches) were taken using the Barco Demetra after technical issues arose that prohibited the continued use of the Dermlite Cam.
Procedure: Skin biopsy — A skin biopsy is a small procedure that removes a sample of skin from the surface of the body. The method utilized will be either a shave or punch technique. The maximum size of a punch biopsy will be 6mm and these wounds are generally closed with no more than 2-3 sutures. A skin biopsy takes <15 minutes including preparation time, administration of intradermal anesthesia using lidocaine 1% with epinephrine 1:100,000, removal of the skin sample, achievement of hemostasis, dressing the wound, and providing instructions for home care. Samples will be placed formalin for routine processing.
Device: Barco Demetra — Barco Demetra is a non-invasive skin imaging system, which acquires multispectral and white light dermoscopic images and clinical photographs of the skin which can then be stored, retrieved, displayed, and reviewed by medical practitioners. The Barco Demetra received 510(k) Premarket approval (K192829). The system involves a hardware imaging device and a stand-alone software application. The hardware device is a portable, battery-powered medical device for acquiring and visualizing images of the skin and uploads all images to cloud storage. The software application is cloud software with an associated web application; it can be used to visualize images and related data and can generate consultation reports. For the purposes of this study, teledermatology images (dermoscopic and clinical - at approximately 6 inches, 12 inches, and 18 inches) were taken using the Barco Demetra after technical issues arose that prohibited the continued use of the Dermlite Cam.

SUMMARY:
The overall goal of this research is to develop a platform that can increase patient access to expert skin cancer diagnostic services via telemedicine. This is especially important for medically underserved areas where melanoma outcomes are worse than in areas with greater access to in-person evaluations. If successful, the widespread availability of such services would be combined with public education efforts to encourage individuals with changing skin lesions to seek evaluation. With decreased travel times to high quality diagnostic services, such efforts may decrease the diagnosis of more advanced melanomas (with a concomitant increase in the diagnosis of earlier stage tumors), and potentially decrease melanoma mortality.

DETAILED DESCRIPTION:
This is a prospective pilot study of a store-and-forward telemedicine diagnostic assessment of participant-selected skin lesions concerning for skin cancer, controlled against an in-person dermatologist assessment (gold standard evaluation). The study will be a single arm design with each participant undergoing telemedicine data acquisition (i.e. clinical and dermoscopic imaging and Nevisense measurement), immediately followed by the in-person dermatologist assessment. The in-person dermatologist will be blinded to the Nevisense score at the time of the visit. Using the telemedicine data, the teledermatology team will render a biopsy/no-biopsy recommendation within 3 business days of the participant evaluation. They will be blinded to the results of the in-person dermatologist's diagnostic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Have 1-3 lesions for evaluation

Exclusion Criteria:

* Lesions of the hair-bearing scalp, in the mouth, on the lips, genitalia, nails, on/around the eyes, inside the ear

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Polsky, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to David.Polsky@nyulangone.org To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Skin lesions
Period: Overall Study
Arm/Group | Participants With Skin Lesions
Started | 149; 378 Skin lesions
Participants Completed Telemedicine Evaluation Visit | 148; 377 Skin lesions
Participants Completed In-Person Evaluation Visit | 148; 377 Skin lesions
Completed | 147; 375 Skin lesions
Not Completed | 2; 3 Skin lesions
Not completed — Screen failure | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Age, Continuous [Median (Full Range); unit: years] | 65 [23 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 121
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 22
  White | 103
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  United States | 147

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Skin Cancer Diagnosis: In-Person Assessment
Description: To compare the accuracy of skin cancer diagnoses between in-person recommendation and the telemedicine (tele) recommendation, the number of "positive" evaluations (i.e. recommended for biopsy) that were truly skin cancer plus the number of "negative" evaluations (i.e. not recommended for biopsy) that were truly non-cancerous divided by the total number of skin lesions evaluated is calculated.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (skin lesions) | 375
percentage of skin lesions | 93 [90 to 95]

2. Primary Outcome: Accuracy of Skin Cancer Diagnosis: Telemedicine Without Nevisense
Description: as for outcome 1
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (skin lesions) | 375
percentage of skin lesions | 91 [88 to 93]

3. Primary Outcome: Accuracy of Skin Cancer Diagnosis: Telemedicine With Nevisense
Description: as for outcome 1
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (skin lesions) | 375
percentage of skin lesions | 83 [79 to 87]

4. Secondary Outcome: Sensitivity of Telemedicine Evaluation in Diagnosing Skin Cancer: Without Nevisense
Description: Assessment of the dermatologist's ability to designate an individual who has skin cancer as "positive" using the telemedicine platform without nevisense.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 85 [57 to 97]

5. Secondary Outcome: Sensitivity of Telemedicine Evaluation in Diagnosing Skin Cancer: With Nevisense
Description: Assessment of the dermatologist's ability to designate an individual who has skin cancer as "positive" using the telemedicine platform with nevisense.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 92 [65 to 100]

6. Secondary Outcome: Sensitivity of In-Person Evaluation in Diagnosing Skin Cancer
Description: Assessment of the dermatologist's ability to designate an individual who has skin cancer as "positive" during in-person evaluations.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 85 [57 to 97]

7. Secondary Outcome: Specificity of Telemedicine Evaluation in Diagnosing Skin Cancer: Without Nevisense
Description: Assessment of the dermatologist's ability to designate an individual who does not have skin cancer as "negative" using the telemedicine platform without nevisense.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 91 [88 to 94]

8. Secondary Outcome: Specificity of Telemedicine Evaluation in Diagnosing Skin Cancer: With Nevisense
Description: Assessment of the dermatologist's ability to designate an individual who does not have skin cancer as "negative" using the telemedicine platform with Nevisense.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 83 [79 to 86]

9. Secondary Outcome: Specificity of In-Person Evaluation in Diagnosing Skin Cancer
Description: Assessment of the dermatologist's ability to designate an individual who does not have skin cancer as "negative" during in-person evaluations.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 93 [90 to 95]

10. Secondary Outcome: False-Positive Rate of Telemedicine Evaluation: Without Nevisense
Description: The number of false-positives (i.e., diagnosing a patient with skin cancer when no skin cancer is present) out of the total number of telemedicine evaluations without Nevisense.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 9 [6 to 12]

11. Secondary Outcome: False-Positive Rate of Telemedicine Evaluation: With Nevisense
Description: The number of false-positives (i.e., diagnosing a patient with skin cancer when no skin cancer is present) out of the total number of telemedicine evaluations with Nevisense.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 17 [13 to 21]

12. Secondary Outcome: False-Positive Rate of In-Person Evaluation
Description: The number of false-positives (i.e., diagnosing a patient with skin cancer when no skin cancer is present) out of the total number of in-person evaluations.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 7 [5 to 10]

13. Secondary Outcome: False-Negative Rate of Telemedicine Evaluation: Without Nevisense
Description: The number of false-negatives (i.e., indicating a patient does not have skin cancer when skin cancer is present) out of the total number of telemedicine evaluations without Nevisense.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 1 [0 to 2]

14. Secondary Outcome: False-Negative Rate of Telemedicine Evaluation: With Nevisense
Description: The number of false-negatives (i.e., indicating a patient does not have skin cancer when skin cancer is present) out of the total number of telemedicine evaluations with Nevisense.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 0 [0 to 2]

15. Secondary Outcome: False-Negative Rate of In-Person Evaluation
Description: The number of false-negatives (i.e., indicating a patient does not have skin cancer when skin cancer is present) out of the total number of in-person evaluations.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 1 [0 to 2]

16. Secondary Outcome: Positive Predictive Value of Telemedicine Evaluation: Without Nevisense
Description: The probability that a patient with a positive (abnormal) test result via telemedicine evaluation without Nevisense actually has skin cancer.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 26 [15 to 40]

17. Secondary Outcome: Positive Predictive Value of Telemedicine Evaluation: With Nevisense
Description: The probability that a patient with a positive (abnormal) test result via telemedicine evaluation with Nevisense actually has skin cancer.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 16 [9 to 26]

18. Secondary Outcome: Positive Predictive Value of In-Person Evaluation
Description: The probability that a patient with a positive (abnormal) test result via in-person evaluation actually has skin cancer.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 31 [18 to 47]

19. Secondary Outcome: Negative Predictive Value of Telemedicine Evaluation: Without Nevisense
Description: The probability that a person with a negative (normal) test result via telemedicine evaluation without Nevisense is truly free of disease.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 99 [98 to 100]

20. Secondary Outcome: Negative Predictive Value of Telemedicine Evaluation: With Nevisense
Description: The probability that a person with a negative (normal) test result via telemedicine evaluation with Nevisense is truly free of disease.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 100 [98 to 100]

21. Secondary Outcome: Negative Predictive Value of In-Person Evaluation
Description: The probability that a person with a negative (normal) test result via in-person evaluation is truly free of disease.
Time Frame: End of the study (4 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of skin lesions
Units Other Than Participants: Skin lesions
Arm/Group | Participants With Skin Lesions
Number analyzed (Participants) | 147
Number analyzed (Skin lesions) | 375
percentage of skin lesions | 99 [98 to 100]

ADVERSE EVENTS:
Time Frame: 4 months
Description: Non-systematic - patient self-report
Arm/Group | Participants With Skin Lesions
All-Cause Mortality (participants affected / at risk) | 0/147
Serious Adverse Events (participants affected / at risk) | 0/147
Other Adverse Events (participants affected / at risk) | 1/147
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Skin Lesions (N=147)
Minor skin infection (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT04411810/Prot_SAP_000.pdf